CLINICAL TRIAL: NCT00037492
Title: Psychological Intervention in Stroke Recovery
Brief Title: Families In Recovery From Stroke Trial (F.I.R.S.T.)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: R01NS032324 (NIH)
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Stroke
Keywords: stroke; recovery
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Procedure: home-based sessions/family meetings with trained clinician

SUMMARY:
The purpose of this trial is to assess the effects of a psychosocial intervention on functional recovery after stroke.

DETAILED DESCRIPTION:
Prior research shows that, after a stroke, emotional support from friends and family is very important in recovery from stroke. This study was designed to test whether a program of family sessions would lead to a faster recovery for stroke patients and lower stress for their families. The sessions were designed to mobilize the family and close friends of a stroke patient and help them to provide effective support to the patient. The aim of the study was to help patients who have recently had a stroke to achieve greater functional ability. Participants were randomly assigned to either the standard care or the treatment group. Those in the treatment group received standard care plus a maximum of 16 home-based sessions, or family meetings, with a specially-trained clinician. (The majority of participants received 14 or 15 sessions.) The sessions included stroke education, information about services and community resources, assistance with problem solving to aid in gaining independence, help with coping, and emotional support. The study is no longer enrolling patients and the study data has been collected. The data is now being analyzed.

ELIGIBILITY:
Inclusion:

* patients with ischemic stroke or non-traumatic intracerebral hemorrhage, with residual deficit origin;
* age 45 or older
* stroke severity (3-8 on the NIH stroke severity scale); and
* able to participate in the intervention (due to, for example, ability to communicate or level of social connectedness).

Exclusion:

* patients living outside the greater Boston area;
* admitted from a nursing home;
* terminally ill;
* severely aphasic;
* significantly cognitively impaired;
* unable to speak English; and
* under 45 years of age.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Berkman, PhD, Principal Investigator — Harvard School of Public Health, Department of Society, Human Development, and Health
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Youville Rehabilitation Hospital, Cambridge, Massachusetts
  - Mount Auburn Hospital, Cambridge, Massachusetts